CLINICAL TRIAL: NCT03605602
Title: TRUMPRWS: A Non-interventional Study on Genetic Variants and Its Clinical Relevance in Chinese Patients With Advanced NSCLC (TRUMPRWS)
Brief Title: A Real World Study Based on NGS (TRUMPRWS)
Acronym: TRUMPRWS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1705
Record Dates: First submitted 2018-07-05; First posted 2018-07-30 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Non-Small Cell Carcinoma of Lung, TNM Stage 4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No treatment is included in this protocol. — No drug intervention or tissue sampling will be included in this study.

SUMMARY:
This is a descriptive observational study, in which data are collected in an epidemiological fashion. This study does not intend to alter or intervene the current medical practice of the recruited patients. Data will be collected in prospective manner.

DETAILED DESCRIPTION:
This is a descriptive observational study, in which data are collected in an epidemiological fashion. This study does not intend to alter or intervene the current medical practice of the recruited patients. Data will be collected in prospective manner.

The eligible patients will be recruited after NGS analysis for tumor tissue and the inform-consent is obtained. The study required information will be collected (every 3 months).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥20 years of age.
2. Provision of fully informed consent prior to any study specific procedures.
3. Histologically or cytologically confirmed, unresectable stage IIIB or stage IV NSCLC.
4. Genetic variants of tumor tissue detected by NGS.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical relevance between genomic profiling and overall survival | [ Time Frame: From registration onto that step until death, or censored at the date of last contact, assessed up to 3 years]
  Kaplan-meier analysis of overall survival based on different genetic alteration

SECONDARY OUTCOMES:
The characteristics of genomic variation and dynamic changes during different anti-tumor treatment | 24 months
  Subtypes, incidence and dynamic changes of genomic variants during treatment process.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, Professor, Study Chair — Guangdong Association of Clinical Trials (GACT)
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, School of Medicine, South China University of Technology, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu SM, Tu HY, Wei XW, Yan HH, Dong XR, Cui JW, Zhou Z, Xu CR, Zheng MY, Li YS, Wang Z, Bai XY, Li AN, Sun YL, Huang J, Lin JX, Ke EE, Xu BF, Lu C, Du Y, Chen Y, Ma R, Wang BH, Cang SD, Wang BC, Chen HJ, Yang JJ, Li Y, Zhou Q, Wu YL. First-line pyrotinib in advanced HER2-mutant non-small-cell lung cancer: a patient-centric phase 2 trial. Nat Med. 2023 Aug;29(8):2079-2086. doi: 10.1038/s41591-023-02461-x. Epub 2023 Jul 24. PMID 37488286
- [Derived] Liu SM, Yan HH, Wei XW, Lu C, Dong XR, Du Y, Cui JW, Chen Y, Ma R, Wang BH, Zhou Z, Cang SD, Yang JJ, Tu HY, Zhang XC, Zhong WZ, Zhou Q, Wu YL. Biomarker-Driven Studies With Multi-targets and Multi-drugs by Next-Generation Sequencing for Patients With Non-Small-Cell Lung Cancer: An Open-Label, Multi-center, Phase II Adaptive Umbrella Trial and a Real-World Observational Study (CTONG1702&CTONG1705). Clin Lung Cancer. 2022 Nov;23(7):e395-e399. doi: 10.1016/j.cllc.2022.05.009. Epub 2022 May 11. PMID 35659479